CLINICAL TRIAL: NCT01376375
Title: A Pilot Study to Evaluate the Effect of Acupuncture on Epigenetic Regulation of Inflammatory Mediators in Participants With Chronic Low Back Pain
Brief Title: Acupuncture to Reduce Signs of Inflammation in Participants With Chronic Low Back Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Purpose: Treatment
Other Study IDs: 110188; 11-AT-0188
Record Dates: First submitted 2011-06-17; First posted 2011-06-20 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2013-04-26

CONDITIONS: Pain
Keywords: Acupuncture; Low Back Pain
MeSH Terms: conditions — Pain; Low Back Pain | interventions — Acupuncture Therapy

INTERVENTIONS:
Procedure: Acupuncture

SUMMARY:
Background:

- Acupuncture is a traditional Chinese medical treatment. Thin needles are used to stimulate specific points in the body. Previous studies have found that acupuncture can be useful in treating low back pain. This study will explore how acupuncture affects low back pain. Researchers will look at blood samples for changes in different chemicals related to inflammation and pain.

Objectives:

- To test the effect of acupuncture on blood chemicals associated with chronic low back pain.

Eligibility:

* People at least 18 years of age who have chronic low back pain.
* Those who have had back surgery or had acupuncture for any medical condition may not participate.

Design:

* This study requires eight visits over 2 to 3 weeks. Each visit will take 1.5 to 2 hours.
* At the first study visit, participants will give a medical history and complete two questionnaires about their low back pain. They will also spend 30 minutes lying down on a bed, relaxing quietly.
* The next visits will occur every 2 to 3 days for the next 2 weeks. Participants will receive 30 minutes of either sham or standard acupuncture. Sham acupuncture will mimic the standard procedure, but no needles will be used. The standard procedure will be performed in the same location. A licensed, experienced acupuncturist will insert small disposable needles into acupuncture sites on the back, arms, and legs. Those in the study will not know whether they are receiving the sham or the standard acupuncture procedure.
* At some visits, participants will provide blood samples for testing. At every visit, participants will complete the questionnaires about low back pain.

DETAILED DESCRIPTION:
Objective:

Inflammation and primary mechanical derangements are thought to be the two major causes leading to low back pain (LBP) syndromes. Increasing evidence suggests that cytokines and hormones, including IFN-gamma, IL-17, IL-1beta, IL-6, TNF-alpha, MMP10, NGF, PGE2, NO and IL-8, play critical roles in the pathogenesis of inflammatory LBP. This study will investigate the effect of acupuncture on LBP by measuring serum cytokine and hormone levels before and after treatment in participants. To define the molecular mechanism by which acupuncture affects LBP, histone modification, including H3K4me3 and H3K27me3, as well as methylation patterns of CpG islands on the promoters of selected genes in the peripheral CD4(plus) T cells will be also tested.

Study Population:

Five participants with chronic LBP will receive treatment.

Design:

In this non-randomized, single group pilot study, participants will be given sham acupuncture and subsequently treated with acupuncture for a total of eight visits over the span of 17 days. Blood will be drawn and analyzed at scheduled intervals.

Outcome Measure:

The primary outcome is to investigate the potential effect of acupuncture treatment, as compared to sham acupuncture and quiet relaxation, on the regulation of IFN-gamma and IL-17 in participants with LBP, including the serum level of these two cytokines, frequency of CD4(plus)IFN-gamma(plus) and CD4(plus)IL-17(plus) cells in the peripheral blood, and the patterns of H3K4me3, H3K27me3 and DNA methylation on their promoters in CD4(plus) T cells in response to acupuncture treatment. Secondary outcomes investigate the effects of acupuncture, as compared to sham acupuncture and quiet relaxation, on the following outcome measures: level of serum cytokines and hormones, including IL-1beta, TNF-alpha, MMP10, NGF, PGE2, NO, IL-8, IL-6, TGF-beta, IL-10, IL-22, IL-23 and IL-17F before and after acupuncture treatment; genome-wide gene expression profile of CD4(plus) T cells before and after acupuncture treatment; genome-wide patterns of H3K4me3 and H3K27me3 modification in CD4(plus) T cells before and after acupuncture treatment; genome-wide patterns of H3K4me3 and H3K27me3 modification in CD4(plus)T cells before and after acupuncture treatment; DNA methylation status change of selected CpG islands before and after acupuncture treatment; and the severity of LBP before and after two weeks of acupuncture treatment according to the Brief Pain Inventory-Short Form (BPI-SF) for pain severity, as well as the Randall Morris Disability Questionnaire (RMDQ) for LBP-related interference scores.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participant must be greater than or equal to 18 years of age.
* Participant must understand and sign the protocol s informed consent document.
* Participant must have been diagnosed with chronic LBP between 3-12 months prior to enrollment.
* Participant must have LBP of greater than or equal to 3 points on a scale of 0 to 10 recorded on the BPI-SF at enrollment.
* Participant must have a RMDQ score of greater than or equal to 3.
* Participant must be able to comprehend English in order to complete questionnaires.

EXCLUSION CRITERIA:

* Participant is unable to comply with study procedures or follow-up visits.
* Participant is in another investigational study and actively receiving study therapy for LBP.
* Participant has received prior treatment with acupuncture for any medical conditions.
* Participant used analgesics, such as opiates or tramadol, within 30 days of enrollment.
* Participant has a significant medical or psychiatric condition that would preclude study completion as determined by the investigator.
* Participant has received corticosteroid treatment within 3 months of enrollment.
* Participant is receiving physical therapy, heat therapy, ultrasound, spinal manipulation, cognitive-behavioral therapy, biofeedback or anticonvulsants for his/her LBP.
* Participant has had back surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-06-10; Primary Completion 2013-04-26 (Actual); Study Completion 2013-04-26 (Actual)

PRIMARY OUTCOMES:
To investigate the potential effect of acupuncture treatment on epigenetic regulation of inflammatory factors in participants with BP

CONTACTS AND LOCATIONS:
Overall Officials: Lai Wei, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Lewis K, Abdi S. Acupuncture for lower back pain: a review. Clin J Pain. 2010 Jan;26(1):60-9. doi: 10.1097/AJP.0b013e3181bad71e. PMID 20026956
- [Background] Ross JS. Non-mechanical inflammatory causes of back pain: Current concepts. Skeletal Radiol. 2006 Jul;35(7):485-7. doi: 10.1007/s00256-006-0121-5. No abstract available. PMID 16752161
- [Background] Cuellar JM, Golish SR, Reuter MW, Cuellar VG, Angst MS, Carragee EJ, Yeomans DC, Scuderi GJ. Cytokine evaluation in individuals with low back pain using discographic lavage. Spine J. 2010 Mar;10(3):212-8. doi: 10.1016/j.spinee.2009.12.007. PMID 20207331